CLINICAL TRIAL: NCT07104331
Title: SARC046: A Phase II Trial of Nab-Sirolimus in Patients With Progressing or Symptomatic Epithelioid Hemangioendothelioma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC046
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Epithelioid Hemangioendothelioma (EHE)
MeSH Terms: conditions — Hemangioendothelioma, Epithelioid

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, open label, single arm Phase II trial with a two stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- non-randomized, open label, single arm (Experimental)
  Interventions: Drug: nab-Sirolimus

INTERVENTIONS:
Drug: nab-Sirolimus — nab-Sirolimus 100 mg/m2 will be administered as an intravenous infusion over 30 minutes on Days 1 and 8 of each 21-day cycle.

SUMMARY:
This is a non-randomized, open label, single arm Phase II trial with a two-stage design with histologically-confirmed metastatic and/or recurrent epithelioid hemangioendothelioma requiring systemic treatment. nab-Sirolimus 100 mg/m2 will be administered as an intravenous infusion over 30 minutes on Days 1 and 8 of each 21-day cycle. The primary objective is to determine ORR by RECIST v1.1 of nab-sirolimus in patients with EHE who require systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed EHE that is either progressing or clinically symptomatic, not a candidate for curative intent surgery, and requires systemic therapy in the opinion of the investigator.
* Participants must have measurable disease by RECIST v1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Age ≥18 years
* ECOG performance status ≤2
* Participants must meet the following organ and marrow function as defined below:

  * Platelets >75,000μl
  * ANC >1500μl
  * Hgb >9g/dl
  * Creatinine <1.5 x ULN or measured CrCl of >30ml/m2/1.73 m2
  * Total bilirubin <2 x ULN
  * AST/ALT <3 x ULN
* Patients must have recovered from toxicity related to prior therapy to grade <=1 (defined by CTCAE v5.0) (except alopecia and neuropathy, or immunotherapy related hypothyroidism). Toxicities that are permanent, like hearing loss from platinum agents, may be allowed if agreed to by the medical monitor.
* The effects of nab-sirolimus on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of nab-sirolimus administration.
* Female patient of childbearing potential has a negative serum pregnancy test within 7 days of study enrollment.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged).

Exclusion Criteria:

* Patient with current evidence of active and uncontrolled infection, NYHA Class III-IV CHF, documented Child's class B-C cirrhosis, or uncontrolled medical disease which in the opinion of the investigator or the sponsor could compromise safety and/or assessment of efficacy.
* Active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative PCR result before enrollment; those who are PCR positive will be excluded. HIV+ patients are allowed provided the patient has a CD4 count greater than 200 and is HIV undetectable on antiviral medications, and there are no AIDS-defining illnesses within 12 months. The antiviral medication regimen must not contain a strong CYP3A4 inhibitor (eg protease inhibitors).
* Major surgical procedure or open surgical biopsy within 28 days of first dose of study drug
* Active central nervous system (CNS) disease involvement, or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity. Subjects with known CNS metastases that are treated and stable (without evidence of CNS toxicity) and are not requiring systemic steroids are allowed to be enrolled.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Myocardial infarction within 12 months of screening
* Co-existing malignancies or use of any other concurrent investigational agents or anticancer agents, excluding adjuvant hormonal therapy for breast or prostate cancer.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nab-sirolimus, breastfeeding should be discontinued if the mother is treated with nab-sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | Approximately 24 months
  To determine ORR by RECIST v1.1 of nab-sirolimus in patients with EHE who require systemic treatment.

SECONDARY OUTCOMES:
Progression-free survival | Month 6 and 12
  The time from starting treatment until disease progression
Duration of response | Approximately 12 months
  The time from tumor response to disease progression

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - Sloan Kettering Institute for Cancer Research, New York, New York

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.